CLINICAL TRIAL: NCT03762525
Title: Anatomic Dynamics of the Internal Iliac Artery After Placement of Iliac Branched Devices Using ECG-gated Computer Tomography Angiography Imaging (IBD-dynamics)
Brief Title: Iliac Branch Device Movement During Cardiac Cycle (IBD-dynamics)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, Prof. Dr., Principal Investigator, Rijnstate Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IBD-dynamics
Record Dates: First submitted 2018-10-05; First posted 2018-12-03 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Iliac Aneurysm; Angiography; AAA
MeSH Terms: conditions — Iliac Aneurysm

STUDY DESIGN:
Intervention Model Description: This study is designed as a multicenter prospective case series.
  1. To prospectively enroll 15 patients that are scheduled for endovascular aneurysm repair using the Gore IBE device in conjunction with its dedicated self expanding Internal Iliac component.
  2. Tocompare 15 patients that have been treated in the period October 2006- July 2016 with the Cook IBD with a non-dedicated IIA component (Advanta-V12 or Fluency) and 15 matched patients treated with Gore IBE device.
Masking Description: The choice for the device is not part of this study and will be made by the doctor in consultation with the patient and the patients anatomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECG gated CTA pre and post operative at Gore IBE (Other): To prospectively enroll 15 patients that are scheduled for endovascular aneurysm repair using the Gore IBE device in conjunction with its dedicated self expanding Internal Iliac component. Each patient will have an ECG gated CTA scan before the operation and 6-8 weeks after operation, in stead of a regular CT scan.
  Interventions: Radiation: ECG gated CTA
- ECG gated CTA post operative at Gore IBE and Cook IBD (Other): To compare 15 patients that have been treated in the period October 2006- July 2016 with the Cook IBD with a non-dedicated IIA component (Advanta-V12 or Fluency) and 15 matched patients treated with Gore IBE device. Each patient will have an ECG gated CTA after the operation, at the first doctor's appointment, in stead of a regular CT scan.
  Interventions: Radiation: ECG gated CTA

INTERVENTIONS:
Radiation: ECG gated CTA — Routine care consists of a preoperative and several postoperative CTA scans. In A. The preoperative and first postoperative CTA will be replaced by ECG-gated CTA imaging and in B. the scheduled imaging will be replaced by an ECG-gated CTA.
  General information: The protocol is based on the ECG gated cardiac protocol using abdominal parameter settings.

SUMMARY:
The incidence of isolated common iliac artery (CIA) aneurysms is low, but in combination with an abdominal aortic aneurysm (AAA) they are found in approximately 20-40% of cases. Basically, two different endovascular strategies can be applied to treat a CIA aneurysm with, including 1. the coverage and 2. the preservation of blood flow to the internal iliac artery (IIA). Coil and coverage of the IIA is related to ischemic complications, including buttock claudication, erectile dysfunction and the more severe spinal and colonic ischemia. Iliac branched devices (IBD) have been developed to exclude CIA aneurysms preserving the IIA and currently three alternatives are on the market. Clinical results of these devices are promising but loss of patency is not uncommon. The major difference between the two devices is the IIA component. The Cook IBD uses a -non-dedicated IIA component, while in the GORE® EXCLUDER® Iliac Branch Endoprosthesis (Gore IBE device) a dedicated self expanding stent is used. Stresses and forces exerted onto the endograft by aortic pulsatility may have an effect on the durability and functioning of the endograft. Intermittent hinchpoints could also have an effect on stent integrity and stenosis. By evaluating endograft movement during the cardiac cycle (ECG-gated CTA) it is possible to assess the stress and force exerted onto the endograft. This might help gain insight into mechanisms underlying potential endograft failure, and aid procedural planning and the development of future devices with long-term durability.

The choice for device is not part of this study.

DETAILED DESCRIPTION:
Objectives:To compare the mobility of the hypogastic artery during the cardiac cycle before and six weeks after implantation of the Gore IBE device in conjunction with its dedicated self expandable Internal Iliac component (Sub-study A);and to quantitatively characterize the displacement of stents with regard to the main body and native IIA during the cardiac cycle on an implanted iliac branched endograft in conjunction with a non-dedicated IIA component (Cook IBD with Advanta V12 or Fluency) with those in conjunction with a dedicated self expandable Internal Iliac component (Gore IBE device). (Sub-study B) Study design: Sub-study A & B: Multicenter observational case studies Study population: Sub-study A: 15 prospectively included patients and sub-study B: 15 patients in each group that have been treated in the period October 2006 - July 2016.

ELIGIBILITY:
Inclusion Criteria:

* Sub-study A. scheduled endovascular aneurysm repair using the Gore IBE device.
* Sub-study B. Patients that have been treated with an iliac branched device in the past in conjunction with either a dedicated IIA component (Gore IBE device) or non-dedicated IIA component (Cook IBD) and who are scheduled for follow-up imaging within the period July 2016-January 2017.

Exclusion Criteria:

* No specific exclusion criteria. Patients will be treated according to the hospital's standard practice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mobility of hypogastric artery during cardiac cycle (sub study A) | Up to 1 year follow-up
  The mobility of the hypogastic artery during the cardiac cycle before and after implantation of the Gore IBE device (Sub-study A). This will be measured at 15 patients by making an ECG gated CTA per and postoperative.
Characterize displacement during cardiac cycle (Sub Study B) | Up to 1 year follow-up
  To quantitatively characterize the displacement during the cardiac cycle on an implanted iliac branched endograft in conjunction with a non-dedicated n balloon expandable IIA component (Cook IBD with Advanta V12 or Fluency) with those in conjunction with a dedicated self expandable Internal Iliac cComponent (Gore IBE device). (Sub-study B). This will be measured by 30 patients (15 pt Cook IBD and 15 pt Gore IBE) an ECG gated CTA postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, MD, PhD, Principal Investigator — Principal Investigator
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem
  - Universitair Medisch Centrum Groningen, Groningen
  - Elisabeth Tweesteden ziekenhuis, Tilburg

IPD SHARING:
Plan to Share IPD: No